CLINICAL TRIAL: NCT06065787
Title: Impact of Peripheral Sensory Stimulation of the Hand and Synchronized Deep Breathing in the Treatment of Anxiety and Depression: Assessing Safety and Effectiveness
Brief Title: NeuroGlove Anxiety and Depression Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NeuroGlove LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REG-1006
Record Dates: First submitted 2023-09-15; First posted 2023-10-04 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Anxiety; Depression; Anxiety Depression; Depression, Anxiety
Keywords: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- NeuroGlove Treatment Arm (Experimental): Subjects will receive treatment using the NeuroGlove. The treatment regimen at home will include 1 hour of therapy per day (two 30-minute sessions, one using each hand) for 4 weeks.
  Interventions: Device: NeuroGlove

INTERVENTIONS:
Device: NeuroGlove — The NeuroGlove is intended to provide peripheral sensory stimulation to the hand through pneumatic puffs of air to encourage collateral blood supply and sensorimotor development.

SUMMARY:
This is a prospective, homebased, interventional clinical study containing 10 subjects who will be enrolled. Approximately 10 (10) subjects with active anxiety and depression symptoms will receive treatment using the NeuroGlove.

DETAILED DESCRIPTION:
This is a prospective, homebased, interventional clinical study containing 10 subjects who will be enrolled. Approximately 10 (10) subjects with active anxiety and depression symptoms will receive treatment using the NeuroGlove.

Subjects will be recruited in from the community. Inclusion in the study will not impact the care management of the subject. Informed consent will be obtained from all subjects before inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* Able to and willing to provide informed consent. Legally authorized representatives (LARs) will not be allowed to consent on behalf of the subject.
* Men and women ≥18 and <85 years of age.
* Carry an active diagnosis of anxiety and/or depression.
* Suffer from anxiety and/or depression symptoms that impact subject's daily activities and quality of life.

Exclusion Criteria:

* Physical limitations of the upper extremity (e.g., fracture, joint deformity, severe spasticity/contracture, wounds, skin breakdown, lymphedema, etc.)
* The subject lacks the ability to comprehend or following instructions, or for any reason, in the opinion of the investigator, would be unlikely or unable to comply with study protocol requirements.
* Currently participating in another interventional clinical trial. (Observational clinical trial participation is allowed for study enrollment.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety symptoms using GAD-7 | 4 weeks
  The change in symptoms pertaining to anxiety will be evaluated using the change in the GAD-7 score. The GAD-7 is a general anxiety questionnaire with 7 questions. The score ranges from 0 - no anxiety to 21 - severe anxiety.
Change in depression symptoms using PHQ-9 | 4 weeks
  The change in symptoms pertaining to depression will be evaluated using the change in the PHQ-9 score. The PHQ-9 is a general anxiety questionnaire with 9 questions. What does a PHQ-9 score mean? Scores less than 5 often signify the absence of a depressive disorder; scores of 5 to 9 predominantly represented patients with either no depression; depression scores of 10 to 14 represented a spectrum of patients; and scores of 15 or greater usually indicated major depression.
Rate of Adverse Events | 4 weeks
  Rate and severity of adverse events related to the use of the NeuroGlove assessed by PI during patient interview.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Nussbaum, MD, Principal Investigator — NeuroGlove LLC
Locations (1):
- NeuroGlove, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with researchers outside of the study. Participant data will be deidentified.